CLINICAL TRIAL: NCT03159559
Title: A Randomized, Open-label Single-center Trial of Lipo-prostaglandin E1 Improves Coronary Microcirculation Dysfunction in Patients With Ischemic Heart Disease Combine With Diabetes Mellitus
Brief Title: PGE1 Improves Coronary Microcirculation Dysfunction in Patients With CAD and Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Chair of Internal medicine Dept. and Cardiovascular Division, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJH-CV-Lipo-PGE1-1
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Coronary Microvascular Perfusion in Patients With Ischemic Heart Disease
MeSH Terms: interventions — Alprostadil; Aspirin; Clopidogrel; Hypoglycemic Agents

ARMS (2):
- Treatment group (Experimental): In the treatment group ,patients received conventional therapy plus Lipo-PGE1 10μg once daily intravenous injection for 7 days ;
  Interventions: Drug: Lipo-PGE1
- Control group (No Intervention): In the control group, patients received conventional therapy only.

INTERVENTIONS:
Drug: Lipo-PGE1 — Patients received conventional therapy plus Lipo-PGE1 10μg once daily intravenous injection for 7 days
  Other Names: aspirin; clopidogrel; antidiabetic drugs
  Arms: Treatment group

SUMMARY:
This study is undertaken to determine if intravenous Lipo-PGE1 therapy would improve coronary microvascular perfusion in patients with ischemic heart disease by CMRI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients giving written consent after being provided with sufficient explanation about participation in this clinical trial
2. Patients aged between 35-70, no limitation on gender
3. Patients with significant CAD and no need to PCI: 50%-70% luminal stenosis as determined by diagnostic coronary angiography, and left main coronary artery stenosis less than 50%; no history of revascularization procedures before
4. MPRI<2.0
5. Type 2 DM patients with glycosylated hemoglobin levels>7%
6. All patients were PGE1-naive, defined as receiving no PGE1 therapy for more than 7 days during the previous 12 months
7. Hypertension remained stable for last 3 months, patients with controlled BP level: SBP<160mmHg and DBP<95mmHg

Exclusion Criteria:

1. Patients with a history of allergic to PGE1 or a history of prior PGE1 treatment.
2. History of revascularization procedures before: PCI or CABG
3. Patients with implanted pacemaker or ICD, ventricular assist device and intra-aortic balloon counter pulsation pump
4. Patients who have experienced myocardial infarction
5. Patients with serious systolic left ventricular function failure: echocardiography EF<25%
6. Claustrophobia
7. Patients who used Insulin pumps
8. SBP<90mmHg
9. Chronic renal function failure: creatinine level >2.5mg/dl or 221umol/l
10. Patients with serious or frequent arrhythmia ,atrial fibrillation、frequent ventricular premature contraction、sick sinus syndrome, second- or third degree atrioventricular block
11. Prior non-cardiac illness with estimated life expectancy <2-yrs
12. Women who are pregnant, lactation,or maybe pregnant in the study period
13. Unable to give informed consent

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
myocardial perfusion reserve index (MPRI) | 1 week